CLINICAL TRIAL: NCT01514357
Title: Novel Peptides in Resistant Human Hypertension
Brief Title: Nesiritide in Resistant Hypertension
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Original PI left the institution, and lack of funding.
Sponsor: John C Burnett (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, John C Burnett, Professor of Medicine and Physiology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-001372; UL1RR024150 (NIH)
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Natriuretic Peptide, Brain; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nesiritide (BNP) (Other): Subjects will receive subcutaneous (SQ) BNP bid for seven consecutive days. The initial starting dose was 5 micrograms/kg.
  Interventions: Drug: Nesiritide (BNP)
- Placebo (Placebo Comparator): Subjects will receive SQ placebo bid for seven consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nesiritide (BNP) — NATRECOR® (nesiritide) is a sterile, purified preparation of human B-type natriuretic peptide (hBNP), and is manufactured from E. coli using recombinant DNA technology. Each 1.5 mg vial contains a white- to off-white lyophilized powder for intravenous (IV) administration after reconstitution.
  Other Names: Natrecor
  Arms: Nesiritide (BNP)
Drug: Placebo — Placebo will be administered subcutaneously instead of active drug (nesiritide) in a blind fashion in the second arm of the study.
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
Hypothesis: If the use of B-type natriuretic peptide (BNP) is proven to be effective in controlling high blood pressure, it may lead to a reduction of standard therapy and improved cardiovascular and kidney protection.

DETAILED DESCRIPTION:
Hypertension remains a global burden in cardiovascular disease leading to stroke, myocardial infarction, and heart failure. Its myocardial complications result from increased mechanical load on the heart. Under physiological conditions of increased myocardial load and resulting myocardial stretch, atrial natriuretic peptide (ANP) and B-type natriuretic peptide (BNP) synthesis and secretion occur contributing to maintenance of optimal cardiorenal and blood pressure homeostasis. However, studies indicate that in subjects with cardiovascular diseases the biological structure of these hormones may be altered, thus reducing their favorable protective activities. New studies indicate that early and moderate hypertension is associated with a derangement of the natriuretic peptide system which is characterized by the lack of activation of biologically active ANP and BNP, while severe hypertension is characterized by cardiac release of altered molecular forms of ANP and BNP that have reduced biological properties and/or enhanced degradation.

The broad objective of proposal is to advance the biology and therapeutics of the natriuretic peptides (NPs) with a special focus on the cardiac peptide BNP in human hypertension. The investigators' proposal is based upon the biological properties of BNP (i.e., natriuretic, renin-angiotensin-aldosterone suppressing, vasodilating, anti-fibrotic, anti-hypertrophic and positive lusitropic), its mechanistic role in human hypertension, and thus its potential as an innovative chronic protein therapeutic to enhance the treatment of patients with uncontrolled and or resistant hypertension. Importantly, BNP is an endocrine hormone normally produced by the human heart, and its use as therapeutic agent has been approved in USA for more than a decade and has been proven to be safe.

ELIGIBILITY:
Inclusion criteria:

Subjects with resistant hypertension as defined by the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC 7) guidelines, systolic blood pressure and/or diastolic blood pressure > 140/90 mm Hg. For patients with hypertension and diabetes or renal disease, blood pressure > 130/80 mm Hg despite treatment with diuretic, sympathetic depressant and vasodilators.

Medications may include a three drug regimen including:

* diuretic at therapeutic dose
* a second line agent such as sympatholytic (e.g. beta-blockade, central agent such as clonidine) or angiotensin converting enzyme inhibitor (ACEi) / angiotensin receptor blocker (ARB) or calcium channel blocker (CCB).
* third line agent including one of the above and/or direct vasodilator, such as hydralazine or minoxidil.

Exclusion criteria:

* Congestive Heart Failure (any New York Heart Association (NYHA) class)
* Ejection Fraction < 50%
* Known renal artery stenosis
* Myocardial infarction within 3 months of screening
* Unstable angina within 14 days of screening, or any evidence of myocardial ischemia
* Moderate to severe pulmonary hypertension
* Valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Sustained Atrial Fibrillation
* Second or third degree atrioventricular (AV) block without a permanent cardiac pacemaker
* Cerebral vascular accident within 3 months of screening, or other evidence of significantly compromised central nervous system perfusion
* Total bilirubin of > 1.5 mg/dL or aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 1.5 times the upper limit of normal range
* Renal insufficiency assessed by calculated Glomerular Filtration Rate (GFR) < 30 ml/min (Cockcroft-Gault equation)
* Serum sodium of < 125 milliequivalent (mEq)/dL or > 160 mEq/dL
* Serum potassium of < 3.0 mEq/dL or > 5.5 mEq/dL
* Women taking hormonal contraceptives
* Pregnancy
* Body mass index (BMI) > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Burnett, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Nesiritide (BNP) | Placebo
Started | 12 | 0
Completed | 8 | 0
Not Completed | 4 | 0
Not completed — Screen failure | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesiritide (BNP) | Placebo | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 0 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in Systolic Blood Pressure (BP)
Description: The change in BP with treatment over 7 days was assessed by the mean BP on admission, (treatment day 1) mean BP 23 hours after the first injection of BNP, and mean BP 23 hours after the second injection of BNP (treatment day 2). Treatment day 2 was 7 days after admission.
Time Frame: baseline, treatment day 1, treatment day 2
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Nesiritide (BNP): Subjects will receive subcutaneous (SQ) Nesiritide (BNP) bid for seven consecutive days. The initial starting dose was 5 micrograms/kg.
Arm/Group | Nesiritide (BNP) | Placebo
Number analyzed (Participants) | 8 | 0
mmHg
  Baseline | 153 (9.180) |
  Treatment Day 1 | 134 (9.07) |
  Treatment Day 2 | 129 (17.34) |

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Nesiritide (BNP) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated early because the original principal investigator left the institution, and also due to the lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes